CLINICAL TRIAL: NCT06596382
Title: A Randomised Double-blind Controlled Trial on Tocotrienol as a Treatment for Non-alcoholic Fatty Liver
Brief Title: Tocotrienol as a Treatment for Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKM PPI/111/8/JEP-2020-190; FF-2020-180 (Other Grant/Funding Number: Sime Darby Oils Nutrition Sdn. Bhd)
Record Dates: First submitted 2023-12-13; First posted 2024-09-19 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Tocotrienol; Vitamin E; Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Intervention Model Description: A randomized double-blinded placebo-controlled trial was performed toward patients diagnosed with NALFD with several established inclusion and exclusion criteria of study. Two main groups were formed to separate the patient into metabolic syndrome and non-metabolic group. In these groups, it will further divided into two groups where the administration of tocotrienol rich-vitamin E and placebo were given in random manner. Each participant will consume the vitamin/placebo daily for one capsule in the duration of six months. Various assessments was conducted before and after taking the vitamin E/placebo.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NAFLD with metabolic syndrome; intervention with tocotrienol rich-vitamin E (Active Comparator): 66 patient diagnosed with NALFD and associated with metabolic syndrome were given 100mg of tocotrienol rich-vitamin E for six months
  Interventions: Dietary Supplement: Tocotrienol rich-vitamin E
- NAFLD without metabolic syndrome; intervention with tocotrienol rich-vitamin E (Active Comparator): 66 patient diagnosed with NALFD without being associated with metabolic syndrome were given 50mg of tocotrienol rich-vitamin E for six months
  Interventions: Dietary Supplement: Tocotrienol rich-vitamin E
- NAFLD with metabolic syndrome; intervention with placebo (Placebo Comparator): 66 patient diagnosed with NALFD and associated with metabolic syndrome were given placebo for six months
  Interventions: Dietary Supplement: Placebo
- NAFLD without metabolic syndrome; intervention with placebo (Placebo Comparator): 66 patient diagnosed with NALFD without being associated with metabolic syndrome were given placebo for six months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tocotrienol rich-vitamin E — Two dosage are available which are 100 mg for NAFLD patient with underlying metabolic syndrome meanwhile 50mg for NALFD patient without metabolic syndrome
  Arms: NAFLD with metabolic syndrome; intervention with tocotrienol rich-vitamin E; NAFLD without metabolic syndrome; intervention with tocotrienol rich-vitamin E
Dietary Supplement: Placebo — Replicate for tocotrienol rich-vitamin E without any active ingredients
  Arms: NAFLD with metabolic syndrome; intervention with placebo; NAFLD without metabolic syndrome; intervention with placebo

SUMMARY:
Vitamin E's potential in treating non-alcoholic fatty liver disease (NAFLD) is attributed to its antioxidant properties. While tocopherols have shown significant results in NAFLD management, the powerful properties of tocotrienols, another form of saturated vitamin E, remain understudied. This research aims to assess tocotrienol's effectiveness in treating NAFLD, expanding our understanding of its therapeutic benefits.

DETAILED DESCRIPTION:
This is a randomized double-blinded placebo-controlled trial targeted toward patients being diagnosed with non-alcoholic fatty liver disease. Patients will be screened and identified from the gastroenterology and hepatology clinic in Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur. The study expects a total of 264 participants to take part in this four-arm investigation, requiring a sample size of 66 for each arm, with an alpha probability of 0.05 and a power of 0.8.

The selection of participants is based on established criteria. The criteria include being 18 years and above, having a high CAP score from FibroScan, and elevated ALT levels. Patients with chronic liver diseases, acute disorders affecting the liver, biliary disease, cancer, and liver cirrhosis were excluded. Alcohol intake was monitored, with a minimum amount set. Any history of bariatric surgery deemed participants unfit for the study. Additionally, participants must be free from the use of steatogenic medication, antibiotics/probiotics, and lipid-lowering agents within one to three months before the study.

After the screening process, participants were assigned to two groups based on metabolic syndrome presence. Within each group, individuals were randomly selected to receive either a vitamin E supplement or a placebo. Each vitamin E capsule contains a certain amount of dosage with a safe concentration for consumption. The metabolic group received 100mg of tocotrienol rich-vitamin E, while the non-metabolic group received 50mg of tocotrienol rich-vitamin E. Meanwhile, each placebo capsule does not contain any vitamin E, which supplied to both group.

Several analyses were performed before and after vitamin E/placebo administration. Firstly, anthropometric data was gathered for their physical measurement. Besides that, FibroScan and LiverFast analysis to examine the liver health condition. Other than that,molecular approach was also conducted to assess the mRNA gene expression level on the selected cytokines such as TNFα, IFNγ, IL-6, and IL-8 and also observe the DNA damage of the cells using Comet Assay. Additionally, biochemical blood testing was tested on 10 parameters to measure its concentration levels within the body. Lastly, each participant was required to answer questionnaires for evaluation on physical activity levels via IPAQ and their dietary patterns through the FFQ

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAFLD is confirmed by the presence of fatty liver detected by abdominal ultrasound and controlled attenuation parameter (CAP) score from FibroScan® of >263 dB/m
* Raised ALT level (above the upper limit of normal): >35 U/L for males and >25 U/L for females

Exclusion Criteria:

* Evidence of other chronic liver diseases (e.g. Hepatitis B, C infections, autoimmune hepatic disorders)
* Evidence of acute disorders affecting the liver (e.g. drug-induced liver injury, non-Hepatitis B, C viral infection)
* Biliary disease
* Liver cancer - primary hepatocellular carcinoma or liver metastasis
* Evidence of liver cirrhosis
* Alcohol intake of >20 g/day for males and 10 g/day for females
* Use of steatogenic medications within the past three months (e.g. systemic steroids, methotrexate)
* History of bariatric surgery
* Intake of antibiotics and/or probiotic supplements within two months prior to the study
* Intake of a lipid-lowering agent (statin) within a month prior to the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Fat percentage before and after intervention in percentage | 6 months
  The measurement were taken using TANITA machine for fat percentage (%) before and after taking vitamin E/Placebo
Fat free mass in kilogram before and after intervention | 6 months
  The measurement were taken using TANITA machine for fat mass, and fat free mass in kilogram, before and after taking vitamin E or Placebo
Basal metabolic rate in kJ before and after intervention | 6 months
  The measurement were taken using TANITA machine for BMR (kJ) before and after taking vitamin E or Placebo
Body Mass Index in kg/m2 before and after intervention | 6 months
  The measurement were taken using TANITA machine for height and weight and will be combined and reported as body mass index (BMI) in kg/m2 before and after taking vitamin E or Placebo
Visceral fat before and after intervention | 6 months
  The measurement were taken using TANITA machine for visceral fat before and after taking vitamin E or Placebo
Liver stiffness based on CAP score before and after intervention | 6 months
  Liver stiffness in the liver was measured using transient elastography technique via FibroScan device, where the evaluation is based on controlled attenuated parameter (CAP) score before and after taking vitamin E/Placebo. CAP score of > 263 indicates fatty liver. The highest score is 1.0. A higher score denotes a worse outcome.
Fatty changes in kPA before and after intervention | 6 months
  Fatty changes in the liver was measured using transient elastography technique via FibroScan device where the evaluation is based on kPA before and after taking vitamin E/Placebo.
Fibrosis via Fibrotest before and after intervention | 6 months
  Blood sample were taken from the patient to determine the degree of liver damage through FibroTest (Fibrosis) based on 10 biomarkers before and after taking vitamin E/Placebo.
Inflammation ActiTest before and after intervention | 6 months
  Blood sample were taken from the patient to determine the degree of liver damage through ActiTest (Inflammation) based on 10 biomarkers before and after taking vitamin E/Placebo.
Steatosis via SteatoTest before and after intervention | 6 months
  Blood sample were taken from the patient to determine the degree of liver damage through SteatoTest (Steatosis) based on 10 biomarkers before and after taking vitamin E/Placebo.
mRNA gene expression level of inflammatory cytokines before and after intervention | 6 months
  Blood sample were taken and extracted for the qualitative determination of mRNA gene expression level of the cytokines (TNFα, IFNγ, IL-6, IL-8) in fold change including housekeeping gene using qPCR method before and after taking vitamin E or Placebo.
DNA damage analysis via Comet assay before and after intervention | 6 months
  Comet assay were conducted to access the DNA damage in the eukaryotic cells via blood sample before and after taking vitamin E/Placebo

SECONDARY OUTCOMES:
Plasma Protein | 6 months
  Protein found in blood which are Alpha-2-macroglobulin, haptoglobin, and apolipoprotein A1 analyzed before and after taking vitamin E/Placebo.
Liver enzymes | 6 months
  Liver enzymes found in blood which are gamma-glutamyl transferase (GGT), alanine transferase (ALT), aspartate aminotransferase (AST) were analyzed before and after taking vitamin E/Placebo.
Triglyceride levels | 6 months
  Triglyceride levels (measured in mg/dL or mmol/L) were analyzed before and after treatment with vitamin E or placebo. Changes in triglyceride levels will be compared to assess the intervention's impact on lipid levels.
Fasting glucose levels | 6 months
  Fasting glucose levels (measured in mg/dL or mmol/L) were analyzed before and after treatment with vitamin E or placebo. Changes in glucose levels will be compared to assess the impact on blood sugar regulation.
Total cholesterol levels | 6 months
  Total cholesterol levels (measured in mg/dL or mmol/L) were analyzed before and after treatment with vitamin E or placebo. Changes in cholesterol levels will be compared to evaluate the effect on lipid metabolism.
International Physical Activity Questionnaire (IPAQ) | 6 months
  Questionnaires related to the physical activity was filled by the patient before and after taking vitamin E or Placebo. The total weekly minutes for each domain will be added up to total the participants' estimated overall physical activity. A longer duration indicates a better outcome.
Food Frequency Questionnaire (FFQ) | 6 months
  Questionnaires related to the food frequency intake was filled by the patient before and after taking vitamin E/Placebo. The food frequency questionnaires give valuable insights into dietary habits by giving out the percentage intake of protein, carbohydrates and total fats. A higher percentage of protein indicates a good diet intake while higher percentages of carbohydrates and total fats indicate a bad diet intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
The investigators are bound to the Institutional Review Board Universiti Kebangsaan Malaysia Medical Research Ethics Committee rules and regulations where recruited patients identity and data are kept confidential and will only be allowed to access by the research team.